CLINICAL TRIAL: NCT00775164
Title: Pioglitazone Therapy in Obese Children With Insulin Resistance: A Randomized, Controlled Pilot Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0811M53986
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obese children with insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pioglitazone (Experimental): Pioglitazone: 15 mg per day for 4 weeks, then up-titrated to 30 mg per day for 12 weeks
  Interventions: Drug: pioglitazone
- Metformin (Active Comparator): Metformin XR; 1000 mg once daily for 16 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: pioglitazone — 15 mg per day for 4 weeks, then up-titrated to 30 mg per day for 12 weeks
  Other Names: ACTOS
  Arms: pioglitazone
Drug: Metformin — Metformin XR; 1000 mg once daily
  Other Names: Glucophage XR
  Arms: Metformin

SUMMARY:
The primary objective of this study is to examine the effects of four months of pioglitazone vs. metformin treatment on HDL cholesterol, triglycerides, blood pressure, insulin resistance, endothelial function, arterial stiffness, adipokines, oxidative stress, and blood biomarkers of endothelial activation in obese insulin resistant children. 30 obese children with elevated fasting insulin levels will be randomly assigned to pioglitazone or metformin for 16 weeks. Change in clinical variables over the 16-week study period will be compared between groups.

DETAILED DESCRIPTION:
Background and Specific Aim/Hypothesis Obese, insulin resistant children are at increased risk of future cardiovascular disease due to elevated systolic blood pressure, fasting insulin, triglycerides, inflammation, oxidative stress, and reduced HDL cholesterol. Behavioral/lifestyle therapy should be the foundational approach to treating obesity and insulin resistance in all individuals, especially children. However, some children may need concomitant medical therapy in order to adequately address their severe risk factor profile and early vascular abnormalities. Although not approved by the FDA, metformin has been used with mixed success to treat obesity-associated cardiometabolic risk factors in children with evidence of insulin resistance. Clearly, other drug therapies should be explored to treat cardiovascular risk factors in obese, insulin resistant children.

Thiazolidinediones have been used to improve glucose control in adult patients with type 2 diabetes mellitus for approximately 10 years. These peroxisome proliferator activated receptor agonists are unique among anti-diabetic agents in that they regulate gene transcription to improve insulin sensitivity in peripheral tissues (predominately skeletal muscle and adipose tissue). In addition to improving glycemic control, these drugs also improve multiple cardiometabolic risk factors such as lipoprotein profile, blood pressure, inflammatory markers, adipokines, and endothelial function. Despite the substantial body of data showing benefit in adults, pioglitazone has never been evaluated as a therapy to improve the cardiometabolic risk factor profile in obese children with evidence of insulin resistance.

Specific Aim: To examine the effects of four months of pioglitazone vs. metformin treatment on HDL cholesterol, triglycerides, blood pressure, insulin resistance, endothelial function, arterial stiffness, adipokines, oxidative stress, and blood biomarkers of endothelial activation in obese, insulin resistant children.

Hypothesis: In the context of background behavioral therapy, four months of pioglitazone vs. metformin treatment will significantly improve HDL cholesterol, triglycerides, blood pressure, insulin resistance, endothelial function, arterial stiffness, adipokines, oxidative stress, and blood biomarkers of endothelial activation in obese insulin resistant children.

Significance There is a substantial lack of data in the literature concerning potential drug therapies for reducing risk factors in children at high risk of developing future cardiovascular disease. Since the prevalence of obesity and insulin resistance in children has increased dramatically in the last several decades, there is an urgent need for data from randomized, controlled trials to guide treatment approaches for high risk children. This pilot study will result in the acquisition of valuable preliminary data which will be used to seek funding for and conduct a larger scale clinical trial evaluating the efficacy of pioglitazone for treating cardiometabolic risk factors in obese, insulin resistant children.

Methods Patient Population: 30 obese, hyperinsulinemic children and adolescents entering a Pediatric Weight Management Program at the University of Minnesota will be enrolled. In this program, children and their families work with a team of trained professionals including physicians, dieticians, and psychologists to reduce weight by making healthier eating choices and increasing physical activity.

Study Design: This will be a randomized, double-blind, active-comparator clinical trial. Variables will be assessed at baseline (prior to randomization) and after four months of therapy.

Data Collection: The screening visit will take place in the Pediatric Weight Management Clinic and will include a complete medical history and physical examination. All research testing will take place in the University of Minnesota General Clinical Research Center (GCRC).

Statistical Analysis and Power Considerations: Randomization will be stratified by gender and Tanner stage. Changes between groups over time will be compared with a 2X2 (group by time) repeated measures ANOVA with Bonferroni post-hoc tests. The main analysis of interest will be the ANOVA interaction term, which compares the change in variables over time (pre vs. post) between groups. The purpose of this study will be to obtain preliminary data to design and seek funding for a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 years old
* Subject able to give assent, and parent/guardian capable of giving consent on behalf of the child
* Body mass index (BMI) ≥ 95th percentile (based on gender and age)
* Fasting insulin ≥ 15 µU/mL AND one or more of the following (cutoffs based on the International Diabetes Federation definition of pediatric metabolic syndrome)1:

  * Triglycerides ≥ 150 mg/dL
  * HDL cholesterol < 40 mg/dL
  * Systolic blood pressure ≥ 130 mmHg

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Has begun a new drug therapy within the past 30 days prior to the screening visit
* BMI ≥ 55
* History of weight loss surgery
* Obesity from a genetic cause (e.g., Prader-Willi)
* Central nervous system injury or severe neurological impairment
* Known systolic or diastolic dysfunction or heart failure
* Females who are currently pregnant or planning to become pregnant
* Liver enzymes > 2.5 times upper limit of normal

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
HDL cholesterol, triglycerides, blood pressure, insulin resistance, endothelial function, arterial stiffness, adipokines, oxidative stress, and blood biomarkers of endothelial activation | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Kelly, Ph.D., Principal Investigator — University of Minnesota